CLINICAL TRIAL: NCT00303173
Title: A Randomized Controlled Trial of The Effectiveness of Guided Imagery on Blood Pressure in Hypertensive Pregnant Women: The Relaxation and Blood Pressure in Pregnancy (REBIP) Pilot Study
Brief Title: The Relaxation and Blood Pressure in Pregnancy (REBIP) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Dalhousie University (Other); AWHONN Canada, with Canadian Nurses Foundation Nursing Care Partnership (Unknown); IWK Health Centre with Canadian Nurses Foundation Nursing Care Partnership (Unknown)
Responsible Party: Faith Wight Moffatt, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16081
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Hypertension; Hypertension, Pregnancy-Induced; Pre-Eclampsia
Keywords: Pre-eclampsia; hypertension; blood pressure; pregnancy; randomized clinical trial; guided imagery; relaxation; psychophysiology; mind-body
MeSH Terms: conditions — Hypertension; Hypertension, Pregnancy-Induced; Pre-Eclampsia | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Guided Imagery

SUMMARY:
Over 10% of women have high blood pressure during their pregnancy which may affect their health or that of their baby. There are currently no methods to prevent most high blood pressure in pregnancy and some treatments are not desirable for use in pregnancy. Previous research indicates that simple relaxation methods can reduce blood pressure and anxiety levels for some people, but this has not been well-studied, especially during pregnancy. This pilot study is intended to determine how guided imagery (imagining relaxing scenes) affects blood pressure and anxiety, and to assess how satisfied women are with this technique. Sixty-six pregnant women with high blood pressure will be randomly assigned to (1) listen to a guided imagery audio-compact disc or (2) quiet rest, at least twice-daily for 4 weeks. All women in both groups will receive all usual care, plus will have their blood pressure measured regularly during 1 day per week for 4 weeks. This study will determine if imagery lowers maternal blood pressure, and if further research on imagery effects on pregnancy health outcomes is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, and less than or equal to (<) 36 weeks, 6 days gestation
* At least two prenatal blood pressure readings > 90 mmHg diastolic
* Has had clinical investigation of the hypertension
* Hearing acuity adequate to hear verbal and audiotaped instructions
* Planning to give birth at one of the study site health centres
* Competent to give informed consent

Exclusion Criteria:

* Likely to deliver within 10 days (including women with diastolic BP >110 mmHg, or systolic BP >170 mmHg; unstable diabetes, concurrent antepartum hemorrhage, preterm labour, and/or other significant medical)
* Prescribed antihypertensive medication at baseline
* Documented psychotic illness
* Unable to understand and read English

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2004-08; Primary Completion 2006-12 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Daytime ambulatory mean arterial pressure | 4 weeks post-randomization (or if delivery is sooner, at most recent ambulatory BP monitoring session

SECONDARY OUTCOMES:
Daytime ambulatory systolic and diastolic blood pressure, and heart rate | 4 weeks post-randomization (or if delivery is sooner, at most recent ambulatory BP monitoring session
Antihypertensive medication use after randomization | between randomization and end of postpartum hospitalization
Maternal anxiety | 4 weeks post-randomization (or if delivery is sooner, at most recent week of available data.
Time to delivery
Relationship of blood pressure changes to reported frequency of guided imagery undertaken
Relationship between classification of hypertension and effectiveness of guided imagery
Relationship between participants' evaluations of their imagery experiences and effectiveness of guided imagery | At 4 weeks post-randomization (or if delivery is sooner, at most recent week od available data)

CONTACTS AND LOCATIONS:
Overall Officials: C. Faith Wight Moffatt, MS, PhD (c), Principal Investigator — University of Toronto, Dalhousie University; Ellen Hodnett, PhD, Study Chair — University of Toronto
Locations (2):
- Canada (2):
  - Womens Health Centre, Eastern Health, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia